CLINICAL TRIAL: NCT06285474
Title: Investigating Low Intensity Focused Ultrasound Pulsation (LIFUP) in Anhedonic Depression
Brief Title: Investigating LIFUP in Anhedonic Depression
Acronym: ILIAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Michelle Craske, Distinguished Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 22-001323
Record Dates: First submitted 2024-02-06; First posted 2024-02-29 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Depression; Anhedonia
Keywords: digital phenotype; ultrasound; depression; anhedonia; imaging
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Caudate (Experimental): Low Intensity Focused Ultrasound Pulsation (LIFUP) will be directed at the caudate head. To minimize the ultrasound energy's exposure to air, a gel pad will be placed between the transducer and the participant's scalp. The sonication protocol will consist of 10 ultrasound sonications in a 30 s ON, 30 s OFF fashion at 650KHz, Ispta≤720 mW/cm2, 50% duty cycle, 5ms pulse width, 1.44W/cm2 ISPPA, and 100Hz pulse repetition frequency." For active sonication, the gel pad will allow the ultrasound energy to pass through. The sham/active gel pads are identical in appearance.
  Interventions: Device: Low Intensity Focused Ultrasound Pulsation (LIFUP)
- Sham Caudate (Sham Comparator): Low Intensity Focused Ultrasound Pulsation (LIFUP) will be directed at the caudate head. To minimize the ultrasound energy's exposure to air, a gel pad will be placed between the transducer and the participant's scalp. The sonication protocol will consist of 10 ultrasound sonications in a 30 s ON, 30 s OFF fashion at 650KHz, Ispta≤720 mW/cm2, 50% duty cycle, 5ms pulse width, 1.44W/cm2 ISPPA, and 100Hz pulse repetition frequency." For sham sonication, the gel pad will block close to all of the ultrasound energy from the transducer from entering the brain. The sham/active gel pads are identical in appearance.
  Interventions: Device: Low Intensity Focused Ultrasound Pulsation (LIFUP)

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound Pulsation (LIFUP) — All participants will undergo 3 identical LIFUP sessions. All sessions must occur at least 1 day apart, and no more than 3 days apart, such that sessions may occur at minimum on days 1, 3, 5 and at maximum may occur on days 1, 5, 9.

SUMMARY:
This study will observe changes in brain imaging, behavior, and symptom measures following intervention with low intensity focused ultrasound pulsation (LIFUP) targeting reward circuitry in individuals who are depressed and anhedonic.

DETAILED DESCRIPTION:
Participants will wear a provided Apple watch and download a study app to their personal phones in order for activity and phone use metrics to be collected. Participants will respond to weekly email surveys, daily ecological momentary assessment (EMA) surveys, complete computer-based neurocognitive assessments, undergo a baseline MRI scan with spectroscopy, receive 3 sessions of LIFUP sonication, undergo a follow up MRI with spectroscopy, then continue to be followed with surveys, neurocognitive assessment, and watch/phone data collection for 3 weeks after follow up MRI scan.

Participants will be randomized 1:1 active:sham to receive LIFUP targeting the caudate head of the brain. Conditions will be double blinded so that neither participants nor investigators or research staff know if active or sham sonication is being administered.

ELIGIBILITY:
Inclusion Criteria:

* • Between the ages of 18 and 65

  * Fluent in English
  * Own functioning iOS smart phone (iPhone 8 or later, iOS 15 or newer) with access to reliable data plan and Wi-Fi
  * Right-handed
  * Normal or corrected to normal vision
  * Willingness to participate in the study, including wearing the provided Apple Watch, respond to remote survey prompts, complete an MRI scan, and provide a recorded interview.
  * Able to read and understand a written informed consent form
  * Reside in the Los Angeles area for the duration of the study
  * If enrolled in IRB#22-000059, have completed the majority of assessments.
  * Eligible for MRI scanning and neuromodulation
  * Willing to receive LIFUP, participate in another MRI scan, keep a study app on their personal phone, and complete 5-7 weeks of assessments.
  * PVSS <6.5 at screening

    * If screened from the general population, PVSS severity must be endorsed in self-report as having lasted for a period of at least 3 months.
    * If screened from IRB#22-000059 scores must average <6.5 at week 6, and stable through study exit. "Stable" defined as the average of all PVSS scores from week 6 through study exit is <6.5
  * PHQ scores > 10 at screening

    * If screened from the general population, PHQ severity must be endorsed in self-report as having lasted for a period of at least 3 months.
    * If screened from IRB#22-000059 scores must average >/= 10 at week 6, and stable through study exit. "Stable" defined as the average of all PHQ scores from week 6 through study exit is >/=10

Exclusion Criteria:

* Current tobacco smoker of >11 cigarettes/day or the nicotine equivalent
* Current report of alcohol or substance abuse or dependence
* Recent changes in antidepressant dosing or medication (dose and medication need to be stabilized within the last 2 weeks)
* Any diagnosis of major neurological condition impairing mobility, cognition, or language ability including multiple sclerosis, Parkinson's disease or other movement disorder, motor neuron disease, stroke, dementia
* Any other diagnosis involving chronic mobility impairment including spinal cord injuries, or severe osteoarthritis of knee or hip
* Reported diagnosis of schizophrenia or psychotic symptoms
* Participants currently taking benzodiazepines must agree to refrain from taking this medication for 12 hours before their scan, as well as refrain from any allergy or cold medication (diphenhydramine) that causes sleepiness (e.g. Benadryl).
* History of brain tumor or brain surgery
* History of stroke or seizure
* Contraindications for MRI scanning, including pregnancy, metal implants, braces, significant grip impairment and claustrophobia
* Unable to complete 3 LIFUP sessions within 1 month of completing the MRI scan for IRB#22-000059
* Unable to complete an MRI scan
* Currently taking benzodiazepines, or taken benzodiazepines in the past 8 weeks
* Any previous treatment with electroconvulsive therapy (ECT) or deep brain stimulation (DBS) due to increased risk of seizure and unclear evidence of how LIFUP will affect individuals who have received these treatments.
* Less than 6 months since any other neuromodulation treatment such as transcranial magnetic stimulation (TMS), Vagal nerve electrostimulation, or transcranial direct current stimulation(TDCS).
* Less than 6 months since prescribed ketamine infusion or other intensive, acute therapy for depressive symptoms.
* History of medical event(s) likely to result in neurological abnormalities including diagnoses of Alzheimer's, Parkinson's, neurodegenerative disorders, movement disorders, or reports of seizures or history of brain tumors.
* Unwilling or unable to refrain from making significant changes to hair style after enrollment and before LIFUP sessions are complete. (ie. full hair style to shaved head, significant change in locs, etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Change in Patient health questionnaire-14 self report measure (PHQ-14) from baseline | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Validated, self-report, 14 item assessment of depressive symptoms in the past 2 weeks. Score range 0- 24. Higher scores indicate higher severity of depressive symptoms.
Change in Positive valence systems scale-21 self report measure (PVSS-21) from baseline | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Validated, self-report 21 item assessment of reward sensitivity. 13 subscales measure different domains of reward sensitivity (range 3-27), with total score (range 1-9) representing overall reward sensitivity. Lower scores indicate more anhedonic responses.
Changes in MRI images from Pre-scan to week 5 | Pre-scan, week 5
  changes in fMRI resting state connectivity, spectroscopy (concentration of glutamate and GABA in the ACC region), and task-based neural activation (using card guessing task) Card Guessing Task: During the scan, participants are asked to guess the value of cards presented on a screen, and are provided immediate feedback as to whether their guesses were correct or not. Participants are informed prior to performing the task, that money is awarded for each correct guess. This task measures reward sensitivity.
  Apple Gathering Task: Effort is expended by participants squeezing a hand-grip measurement tool, which translates a signal to the screen showing the amount of effort they are expending to receive a pre-determined amount of "reward". Participants can accept or reject trials of effort based on the amount of reward they would be due to receive. This task measures reward sensitivity and motivation.
Change in Ecological momentary assessment (EMA) from W0/Baseline | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Ecological momentary assessment (EMA) is a custom 16 item self-report assessment of in-the moment mood and activity. This is a data collection instrument without a standardized scoring method.

SECONDARY OUTCOMES:
Changes in digital behavioral phenotype sleep measurement | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Apple watch & phone sensor metrics of sleep.
Changes in digital behavioral phenotype physical activity measurement | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Apple watch & phone sensor metrics of physical activity.
Changes in heart rate | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Apple watch & phone sensor metrics of heart rate.
Changes in heart rate variability | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Apple watch & phone sensor metrics of heart rate variability.
Changes in respiratory rate | Week 0, Pre-scan, Baseline, week 1, week 2 week 3, week 4, week 5
  Apple watch & phone sensor metrics of respiratory rate.
changes in World Health Organization (WHO) -5 Wellbeing index score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 5 item assessment of self-reported current mental wellbeing. Total score range 0-25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
changes in Pittsburgh Sleep Quality Index (PSQI) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 18 item self-report of recent sleep quality. Domain scores calculate items like sleep latency, disturbance, etc. and are used to calculate total score. Total score range is 0-21 with higher total scores indicating worse sleep quality.

OTHER OUTCOMES:
changes in Quick Inventory of Depressive Symptoms (QIDS-SR15) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 15 item self-report of depressive symptoms. Total score range is 0-24 with higher total scores indicating more severe depressive symptoms.
changes in Patient Health Questionnaire (PHQ-9) score from day 2 to week 2 | Day 2, week 1, week 2
  Validated, self-report 9 item assessment of depressive symptoms including suicidal ideation. Score range 0-27. Higher scores indicate higher severity of depressive symptoms.
changes in Brief Irritability Test (BITe) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 5 item self-report irritability measure. Score range 5-30 with higher scores indicating more irritable responses.
changes in Generalized Anxiety Disorder (GAD-7) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 7 item self-report of anxiety symptoms. Score range 0-21 with higher scores indicating more anxious symptoms.
Changes in Snaith Hamilton Pleasure Scale (SHAPS) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 14 item self-report measure of hedonic experience or positive valence. Total score range is 0-14 with higher scores representing more anhedonic responses.
Changes in Suicidal Ideation measure from Pre-scan to end of study | Pre-scan, week 5
  Custom, 22 item self-report measure of history and current presence of suicidal ideation and behavior. Domain scores assess current and lifetime severity. Score range 0-1 with higher scores indicating more severe suicidal ideation and risk.
changes in Apathy Motivation Index (AMI) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 18 item self-report index of apathy and motivation. Domain scores assess behavioral, social, and emotional responses. Score range for each domain is 0-4 with higher scores indicating more apathetic or unmotivated responses.
changes in Eudaimonic Well-Being Questionnaire (EWBQ) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Custom, 5 item survey assessing self-reported well-being focused on values, meaning and purpose in life. Total score range 0-20 with lower scores reflecting responses of low wellbeing.
Changes in Work and Social Adjustment Scale (WSAS) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 8 item assessment of self-reported functional impairment of current symptoms in work/school, social life, and family life. Total score range 0-40 with higher scores indicating more impairment.
Changes in Ruminative Response Scale (RRS) - brooding subscale score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 9 item assessment of self-reported symptoms of rumination. Total score range 0-27 with higher scores reflecting more rumination.
changes in Trauma History Questionnaire (THQ) score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated self-report measure of traumatic life events. This is a data collection instrument without a standardized scoring method which will be used as a covariate.
changes in Routines Survey from W0/Baseline to end of study | Week 0/Baseline, week 5
  Custom self-report of daily activities and phone usage. This is a data collection instrument without a scoring method.
changes in USDA Housing and Food Insecurity score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 6 item assessment of self-reported household food security. Total score range 0-6 with higher scores indicating higher food insecurity. This measure will be used as a covariate.
changes in Holmes-Rahe Life Stress Survey score from W0/Baseline to end of study | Week 0/Baseline, week 5
  Validated, 40 item assessment of self-reported exposure to moderate-to-major stressful life events. Score range 0-40 with higher scores representing more exposure to stressful life events. This measure will be used as a covariate.
Changes in emotion recognition accuracy scores from Pre-scan to end of study | Pre-scan, week 5
  TestMyBrain is a computer administered neurocognitive battery that will provide scores for emotion recognition accuracy. Where accuracy scores represent the proportion correct responses across trials, with higher scores indicating more accurate responses.
Changes in emotion recognition response times from Pre-scan to end of study | Pre-scan, week 5
  TestMyBrain is a computer administered neurocognitive battery that will provide scores for scores for emotion recognition response times. Higher response times indicate taking longer to generate a response.
Changes in continuous concentration accuracy scores from Pre-scan to end of study | Pre-scan, week 5
  TestMyBrain is a computer administered neurocognitive battery that will provide scores for continuous concentration accuracy. Where accuracy scores represent the proportion correct responses across the trial, with higher scores indicating more accurate responses.
Changes in continuous concentration response times from Pre-scan to end of study | Pre-scan, week 5
  TestMyBrain is a computer administered neurocognitive battery that will provide scores for scores for continuous concentration response times. Higher response times indicate taking longer to generate a response.
Changes in continuous concentration error scores from Pre-scan to end of study | Pre-scan, week 5
  TestMyBrain is a computer administered neurocognitive battery that will provide scores for continuous concentration errors. Error scores represent the proportion errors committed during the trial, with higher scores indicating more errors.
Changes in Apple Gathering task behavior from Pre-scan to end of study | Pre-scan, week 5
  Effort is expended by participants squeezing a hand-grip measurement tool, which translates a signal to the screen showing the amount of effort they are expending to receive a pre-determined amount of "reward". Participants can accept or reject trials of effort based on the amount of reward they would be due to receive. This task measures reward sensitivity and motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected will be deidentified and shared with the team members of this MC Psych research consortium under Wellcome Trust. Shared data types will include individual participant survey responses, self-report diagnostic measures, treatment history, neurocognitive performance, interview data including de-identified face and speech summary metrics, Apple watch metrics, phone usage metrics, fMRI data, demographic data.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data is being made available throughout the course of collection, and will remain available for study for up to 10 years.
Access Criteria: Researchers permitted access to the deidentified data from this study must be a part of the MC Psych consortium, as designated and approved by the sponsor, Wellcome Trust. All other requests for access to data from this project will be reviewed by the principal investigator for approval.